CLINICAL TRIAL: NCT04673812
Title: Influence Of Low Dose Intrathecal Naloxone On Bupivacaine - Fentanyl Spinal Anaesthesia For Lower Limb Orthopedic Surgery In Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, lecturer of anesthesia,SICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS/19.09.830
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia, Spinal; Elderly
Keywords: spinal anesthesia; elderly; naloxone; pruritus; post operative cognitive dysfunction
MeSH Terms: conditions — Pruritus | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine-Fentanyl Spinal Anaesthesia (Active Comparator)
  Interventions: Drug: Bupivacaine-fentanyl
- Bupivacaine-Fentanyl-Naloxone Spinal Anaesthesia (Active Comparator)
  Interventions: Drug: Bupivacaine-fentanyl

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — Bupivacaine-Fentanyl (BF) group (46 patients): will receive spinal anaesthesia with 12.5 mg hyperbaric Bupivacaine 0.5% (2.5 mL) plus 25 µg Fentanyl (0.5 mL) and (0.5 mL) normal saline added in the same syringe in a total volume of 3.5 mL.
  Bupivacaine-Fentanyl-Naloxone (BFN) group (46 patients): will receive spinal anaesthesia with 12.5 mg hyperbaric Bupivacaine 0.5% (2.5 mL) plus 25 µg Fentanyl (0.5 mL) and 20 µg Naloxone (prepared in 0.5 mL normal saline) added in the same syringe in a total volume of 3.5 mL.
  Other Names: Naloxone hydrochloride

SUMMARY:
Fentanyl is a safer alternative than morphine in the management of postoperative pain in elderly. However, pruritus, nausea and vomiting are unwanted side effects of intrathecal fentanyl administration, that can decrease patient satisfaction with anaesthesia, delay post anaesthesia care unit ( PACU ) discharge, and increase costs.

The incidence of pruritus with neuraxial fentanyl is high. The incidence of pruritus in non-obstetric surgery patients after intrathecal fentanyl ranges from 53% to 79%.

Naloxone hydrochloride is a pure opioid competitive antagonist. Small doses of naloxone may reduce Fentanyl-associated adverse effects, such as pruritus, nausea and vomiting without affecting analgesia.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of adding low dose intathecal naloxone to bupivacaine - fentanyl spinal anesthesia in elderly patients scheduled for unilateral lower limb orthopedic surgeries on opioid induced side effects namely pruritus, postoperative analgesia and the incidence of postoperative cognitive dysfunction (POCD) in elderly.

A four category verbal rating scale VRS-4 ( 0 to 3 scale ) will be used for assessment of intrathecal fentanyl induced side effects including pruritus, nausea, vomiting and shivering.

Mini Mental State Examination ( MMSE ) test will be applied to all patients pre- and post- operative to assess the incidence and the degree of POCD.

An 11 points Verbal Numerical Rating Scale VNRS for pain assessment will be also applied to all patients postoperatively to assess the effect on postoperative analgesia.

* Cannulation: Peripheral cannulae ( size 20 gauge or 18 gauge ) will be inserted to all patients . Ringer's acetate warmed up to 37°C will be infused slowly at rate of 7ml/kg, 30 min before induction of spinal anaesthesia. A single intravenous ( I.V. ) dose of prophylactic antibiotic after a negative sensitivity test will be given to all patients 15-30 min. before operation.
* Induction: Patient will receive spinal anaesthesia with 12.5 mg hyperbaric Bupivacaine 0.5% ( 2.5 mL ) plus 25 µg Fentanyl ( 0.5 mL ) and 20 µg Naloxone ( prepared in 0.5 mL normal saline ) added in the same syringe in a total volume of 3.5 mL..
* Spinal anaesthesia will be conducted while the patients are in the sitting position and under complete aseptic conditions; a lumber puncture at L3-4 or L4-5 interspaces will be performed with a 25- gauge Quincke spinal needle after infiltrating the skin with 2 ml of lidocaine 2%. After a successful dural puncture and ensuring free flow of cerebrospinal fluid, injectates will be injected slowly over 20 seconds without barbotage or aspiration according to group of the patient. Immediately, patients will be turned into the supine position. Oxygen 2-3 L/min will be applied to all patients via nasal prongs.

Evolution and regression of sensory and motor block will be evaluated. Sensation will be assessed by pinprick in the mid-clavicular line as follows; Grade 0: Sharp pain felt, Grade I: Analgesia, dull sensation felt, Grade II: Anesthesia, no sensation felt. Motor blockade will be assessed according to Modified Bromage Scale.

Hemodynamics ( mean arterial blood pressure MAP, heart rate HR and oxygen saturation SpO2 ) will be also recorded at predetermined accurate times.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60y of either gender.
* ASA physical status III or below.
* Patients scheduled for elective unilateral lower limb orthopedic surgery.

Exclusion Criteria:

* Morbid obese patients.
* Severe or uncompensated cardiovascular, renal, hepatic or endocrinal diseases.
* Allergy to one of the agents used.
* Severely altered consciousness level.
* Coagulopathy
* Increased intracranial pressure
* Neuromuscular diseases
* Severe spinal deformity
* Patients on opioid analgesics or opioid abuse
* Multi traumatized patients
* Patients with preoperative Mini Mental State Examination ( MMSE ) scoring < 24

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
incidence of fentanyl - induced pruritus | 4 hours postoperative
  A four category verbal rating scale VRS-4 ( 0 to 3 scale ) which will be will be explained to all patients, where ( 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms ) with the basal preoperative value is being recorded.

SECONDARY OUTCOMES:
The time for first postoperative analgesic requirements | 24 hours
Cognitive function using Mini Mental State Examination (MMSE) scoring | 24 hours
postoperative nausea and vomiting | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y. Makharita, professor, Principal Investigator — Mansoura University
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No